CLINICAL TRIAL: NCT05557253
Title: Effects of Remimazolam on the Intraoperative Hemodynamic Parameters in Patients Undergoing Extracranial-intracranial Bypass Surgery: a Prospective Randomized Controlled Trial
Brief Title: Effects of Remimazolam on the Intraoperative Hemodynamics in Bypass Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang-Hoon Koo, Assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Bypass-RMDZ
Record Dates: First submitted 2022-09-25; First posted 2022-09-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Intraoperative Hypotension
MeSH Terms: interventions — remimazolam; Balanced Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remimazolam group (Experimental): General anesthesia is induced and maintained with remimazolam.
  Interventions: Drug: Remimazolam
- balanced group (Active Comparator): General anesthesia is induced with propofol and maintained with desflurane.
  Interventions: Drug: Balanced Anesthesia

INTERVENTIONS:
Drug: Remimazolam — Anesthesia induction: remimazolam 6-12 mg/kg/h Anesthesia maintenance: remimazolam 1-2 mg/kg/h
  Arms: remimazolam group
Drug: Balanced Anesthesia — Anesthesia induction: propofol 1.5-2 mg/kg Anesthesia maintenance: Desflurane 6-8 vol%
  Arms: balanced group

SUMMARY:
This study is a randomized, controlled trial. A total of 72 patients will be randomized to receive remimazolam anesthesia or balanced anesthesia (propofol + desflurane) during extracranial-intracranial bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo elective extracranial-intracranial bypass surgery
* American Society of Anesthesiologists grade 1,2,3
* Age > 18 years old

Exclusion Criteria:

* Refuse to participate to the study
* American Society of Anesthesiologists grade 4
* Body Mass Index < 18.5 kg/m2 or > 35 kg/m2
* Allergic history of benzodiazepine
* Pregnant
* Acute narrow-angle glaucoma
* Shock or Coma
* Acute alcohol addicted
* Obstructive sleep apnea
* dependency on alcohol or drug
* Severe acute respiratory insufficiency
* Hypersensitivity to Dextran 40

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative hypotension | During surgery
  Target Systolic Blood Pressure < 80%

SECONDARY OUTCOMES:
Inotropic requirements | During surgery
  Dose of inotropics administered during surgery
Incidence of bradycardia | During surgery
  heart rate < 40 /min
Incidence of tachycardia | During surgery
  heart rate > 100 /min
Maximum systolic blood pressure | During surgery
  Maximal systolic blood pressure during surgery (mmHg)
Minimum systolic blood pressure | During surgery
  Minimal systolic blood pressure during surgery (mmHg)
Brain relaxation score | Immediately after dura opening
  1=perfectly relaxed, 2=satisfactorily relaxed, 3=firm brain, 4=bulging brain

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hoon Koo, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No